CLINICAL TRIAL: NCT00002506
Title: ALPHA INTERFERON AND CIS-RETINOIC ACID FOR THE TREATMENT OF SQUAMOUS CELL CARCINOMAS
Brief Title: Isotretinoin Plus Interferon in Treating Patients With Recurrent Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Purpose: Treatment
Other Study IDs: CDR0000077957; CBRG-9208; NBSG-9208; NCI-V92-0159
Record Dates: First submitted 1999-11-01; First posted 2004-07-26 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Cervical Cancer; Esophageal Cancer; Head and Neck Cancer; Lung Cancer; Non-melanomatous Skin Cancer; Penile Cancer
Keywords: recurrent non-small cell lung cancer; recurrent esophageal cancer; recurrent cervical cancer; squamous cell lung cancer; squamous cell carcinoma of the skin; recurrent penile cancer; recurrent skin cancer; squamous cell carcinoma of the esophagus; cervical squamous cell carcinoma; penile squamous cell carcinoma; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Penile Neoplasms; Carcinoma, Non-Small-Cell Lung; Skin Neoplasms; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck | interventions — Interferon-alpha; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: isotretinoin

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of isotretinoin may be an effective way to prevent cancer or stop cancer from growing. Interferon alfa may interfere with the growth of cancer cells. Combining isotretinoin and interferon may be an effective treatment for some recurrent cancers.

PURPOSE: Phase II trial to study the effectiveness of interferon alfa plus isotretinoin in treating patients with recurrent cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rates to treatment with daily subcutaneous interferon alpha plus oral isotretinoin in patients with advanced squamous cell carcinomas of the following body sites: head and neck, cervix, skin, esophagus, lung, and penis. II. Determine the toxicities and side effects of this treatment.

OUTLINE: Nonrandomized study. Single-agent Chemotherapy with Biological Response Modifier Therapy. Isotretinoin, 13-CRA, NSC-329481; with Interferon alpha (Schering or Hoffmann-La Roche), IFN-A, NSC-377523 or NSC-367982.

PROJECTED ACCRUAL: 14-50 patients per tumor category (and any other tumor location, if available) will be enrolled. If none of the first 14 patients in any tumor category responds, or if only 1/22, 2/30, 3/37, 4/44, or 5/50 respond, the treatment will be considered ineffective for that tumor type.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma that has failed standard local modalities for local disease and/or effective systemic therapy for metastatic disease, or for which other forms of systemic therapy have been refused Eligible sites include but are not limited to: Uterine cervix Head and neck Skin Esophagus Lung Penis Measurable or evaluable disease required Measurable disease defined as previously unirradiated disease reproducibly measurable in 2 dimensions by physical exam, x-ray, CT, MRI, or other radiologic procedure Documented progressive disease in a previously irradiated site is accepted as measurable Evaluable disease includes: Any visible radiologic disease not measurable in 2 perpendicular diameters Elevated squamous cell carcinoma antigen (SCCA) No active brain metastases Previously treated brain metastases that have responded to therapy do not exclude, but CNS disease is not considered measurable or evaluable

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Hematopoietic: WBC at least 3,000 Platelets at least 100,000 Hct at least 30% Hepatic: Bilirubin less than 2.0 mg/dl PT normal PTT normal Renal: Creatinine less than 2.0 mg/dl Cardiovascular: No MI within 6 months No CHF requiring medication No arrhythmia requiring medication Pulmonary: Reasonable respiratory reserve required No requirement for supplemental oxygen No dyspnea at rest Other: No chronic underlying immunodeficiency disease No HIV positivity No pregnant patients (negative pregnancy test required) Adequate birth control required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No concomitant immunosuppressive drugs, e.g., cyclosporin Chemotherapy: At least 3 weeks since prior systemic chemotherapy with recovery Endocrine therapy: No concomitant corticosteroids Radiotherapy: No prior radiotherapy to measurable site unless disease progression is documented Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-08; Primary Completion 1996-01 (Actual); Study Completion 1999-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (6):
- United States (6):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Bloomington Hospital, Bloomington, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - St. Joseph Regional Cancer Center, Bryan, Texas

REFERENCES:
- [Result] Dillman RO, Soori G, Tai DF, et al.: Interferon alpha-2A (FN) and cis-retinoic acid (CRA) for the treatment of squamous cell carcinoma (SCC): a preliminary report. J Immunother 20(5): 404, 1997.